CLINICAL TRIAL: NCT03557957
Title: Targeted Correction of Plasma Sodium Levels in Hospitalized Patients With Hyponatremia: a Randomized, Controlled, Parallel-group Trial
Brief Title: Targeted Correction of Plasma Sodium Levels in Hospitalized Patients With Hyponatremia
Acronym: HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Erasmus Medical Center (Other); Cantonal Hospital of Aarau, Switzerland (Other); Spital Solothurn, Switzerland (Unknown); Cantonal Hospital of St. Gallen (Other); Kantonsspital Liestal, Switzerland (Unknown); Universitätsklinikum Köln (Other); KBC Zagreb, Croatia (Unknown); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIT-trial
Record Dates: First submitted 2018-05-16; First posted 2018-06-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel-group trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to allocated treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care plus targeted correction of hyponatremia (Experimental): Diagnosis and treatment of hyponatremia will be standardized according to the European Clinical Practice Guidelines (ECPG). Treatment response and adherence will be evaluated daily and treatment adapted if treatment goals are not reached.Targeted correction of plasma sodium Levels.
  Interventions: Other: Targeted correction of plasma sodium levels
- Standard care (Active Comparator): Diagnosis and treatment of hyponatremia will be solely at the discretion of the attending physicians who are in no way involved in the trial. The study team will not intervene with the treatment in any way. Diagnostic and treatment decisions as well as course of the plasma sodium level will only be recorded after patient is discharged from hospital using the medical records and patient charts. It will be generally recommended to measure plasma sodium levels 3x weekly or more frequently if clinically indicated, at discharge and after 30 days.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Targeted correction of plasma sodium levels — Targeted correction of hyponatremia
  Arms: Standard care plus targeted correction of hyponatremia
Other: Standard care — Standard care of hyponatremia
  Arms: Standard care

SUMMARY:
Hyponatremia is the most common electrolyte disorder with a prevalence of up to 30% in hospitalized patients. While treatment of acute hyponatremia with severe clinical symptoms due to cerebral edema is undisputed and straightforward, hyponatremia in general is usually considered asymptomatic or not clinically relevant. Accordingly, a recent observational study showed that appropriate laboratory tests to evaluate the etiology of hyponatremia were obtained in less than 50% of patients, leading to 75% of patients being still hyponatremic at discharge.

This is problematic in the context of increasing evidence, revealing an association of chronic hyponatremia with adverse effects such as gait alterations and falls, attention deficits, bone loss and fractures as well as disease-associated morbidity leading to increased rates of readmissions and mortality. Yet, there is a complete lack of randomized clinical trials with the primary aim to investigate whether correction of plasma sodium concentration counteracts the elevated risk of rehospitalization and mortality.

The aim of this trial is therefore to determine the effects on mortality and rehospitalization rate of a targeted correction of plasma sodium concentration in addition to current standard care in hospitalized hyponatremic patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult hospitalised patients with hypotonic hyponatremia <130mmol/L
* Hospitalization of at least 24 h after inclusion in the study

Exclusion Criteria:

* severe symptomatic hyponatremia in need of intensive care treatment
* non-hypotonic hyponatremia with plasma osmolality >280 milliosmol (mOsm)/kg
* end of life care (palliative treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2278 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the combined risk of death or rehospitalization within 30 days | 30 days
  Rate of death or rehospitalization within 30 days

SECONDARY OUTCOMES:
30 days mortality rate | 30 days
  Mortality rate
1 year mortality rate | 1 year
  Mortality rate
30 days rehospitalization rate | 30 days
  Rehospitalization rate
1 year rehospitalization rate | 1 year
  Rehospitalization rate
Time to rehospitalization | up to 1 year
  Days until first rehospitalization
Time to death | up to 1 year
  Days until death
length of hospital stay | up to 1 year
  length of index hospital stay in days
Rate of falls | 30 days
  Number of falls
Rate of fractures | 30 days
  Number of bone fractures
Rate of fractures | 1 year
  Number of bone fractures
Rate of Plasma sodium normalization at discharge | up to 1 year
  Rate of Plasma sodium Levels >=135mmol/L at discharge
Change in Plasma sodium Levels | up to 1 year
  Change in mmol/L in Plasma sodium Levels from inclusion to discharge
Recurrence of hyponatremia | 30 days
  Rate of recurrence of hyponatremia
Recurrence of hyponatremia | 1 year
  Rate of recurrence of hyponatremia
Severely symptomatic hyponatremia | up to 1 year
  Rate of severely symptomatic hyponatremia requiring intensive care Treatment during index hospitalization
Sodium-overcorrection | up to 1 year
  Rate of plasma sodium overcorrection during index hospitalization
number of adverse events | 30 days
  Rate of adverse events
number of adverse events | 1 year
  Rate of adverse events
Severe adverse events | 30 days
  Rate of severe adverse events
Severe adverse events | 1 year
  Rate of severe adverse events
Diagnostic accuracy of copeptin in the diagnosis of hyponatremia | 1 day
  Copeptin Level will be correlated with final hyponatremia diagnosis
Diagnostic accuracy of mid-regional mid-regional (MR)-proANP in the diagnosis of hyponatremia | 1 day
  MR-proANP Level will be correlated with final hyponatremia diagnosis N-terminal (NT)-proBNP, aldosterone, renin)
Diagnostic accuracy of NT-proBNP in the diagnosis of hyponatremia | 1 day
  NT-proBNP Level will be correlated with final hyponatremia diagnosis
Diagnostic accuracy of aldosterone in the diagnosis of hyponatremia | 1 day
  Aldosterone Level will be correlated with final hyponatremia diagnosis
Diagnostic accuracy of renin in the diagnosis of hyponatremia | 1 day
  Renin Level will be correlated with final hyponatremia diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (9):
- University Hospital Centre Zagreb, Zagreb, Croatia
- Uniklinik Köln, Cologne, Germany
- Careggi University Hospital Florence, Florence, Italy
- Erasmus Medical Center Rotterdam, Rotterdam, Netherlands
- Switzerland (5):
  - University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baselland, Liestal
  - Kantosspital St. Gallen, Sankt Gallen
  - Solothurner Spitäler AG, Solothurn

IPD SHARING:
Plan to Share IPD: Yes
Metadata describing the type, size and content of the datasets will be shared along with the study protocol and case report forms on the public repository dataverse.harvard.edu.
Supporting Information: Study Protocol, ICF, CSR
URL: http://dataverse.harvard.edu

REFERENCES:
- [Derived] Refardt J, Pelouto A, Potasso L, Hoorn EJ, Christ-Crain M. Hyponatremia Intervention Trial (HIT): Study Protocol of a Randomized, Controlled, Parallel-Group Trial With Blinded Outcome Assessment. Front Med (Lausanne). 2021 Sep 6;8:729545. doi: 10.3389/fmed.2021.729545. eCollection 2021. PMID 34552947